CLINICAL TRIAL: NCT07391514
Title: Deep Learning-Based Intraoperative Dual-tracer Video Analysis of Sentinel Lymph Node Mapping for Metastasis Prediction in cN0 Papillary Thyroid Carcinoma: A Prospective Cohort Study
Brief Title: Deep Learning-Based Intraoperative Dual-tracer Video Analysis of Sentinel Lymph Node Mapping for Metastasis Prediction in cN0 Papillary Thyroid Carcinoma
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Xinliang Su, Clinical Professor, First Affiliated Hospital of Chongqing Medical University
Other Study IDs: 1stChongqingMU-sxl
Record Dates: First submitted 2026-01-19; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Papillary Thyroid Carcinoma
Keywords: Papillary thyroid carcinoma; Sentinel lymph node biopsy; Dual-tracer imaging; Indocyanine green; Carbon nanoparticles; Deep learning
MeSH Terms: conditions — Thyroid Cancer, Papillary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Tissue specimens collected during thyroid cancer surgery include:
  1. Sentinel lymph node tissue: The first-draining lymph node identified by dual-tracer mapping, submitted separately for pathological examination.
  2. Central compartment lymph node tissue: Specimens from prelaryngeal, pretracheal, paratracheal regions, and lymph nodes posterior to the recurrent laryngeal nerve.
  3. Lateral compartment lymph node tissue: When indicated based on intraoperative findings.
  4. Thyroid tissue: From lobectomy or thyroidectomy specimens.
  All specimens undergo:
  * Intraoperative frozen section analysis for immediate assessment
  * Postoperative formalin-fixed paraffin-embedded (FFPE) processing for definitive histopathological diagnosis
  * Genetic testing for mutation analysis (including BRAF mutation status)
  Tissue samples are stored according to institutional biobank protocols and may be used for future research with appropriate ethical approval.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ICG Group: Adults with clinically node-negative papillary thyroid carcinoma (cN0-PTC) who undergo intraoperative sentinel lymph node mapping using indocyanine green (ICG) alone.
  Intervention: 0.2 ml of ICG solution (concentration: 2.5 mg/ml) injected at multiple points around the thyroid tumor under ultrasound guidance. Near-infrared fluorescence imaging is used to visualize lymphatic drainage and identify sentinel lymph nodes.
  Participants undergo standard thyroid surgery including thyroid lobectomy and central lymph node dissection, with additional dissection based on intraoperative findings.
  Interventions: Diagnostic Test: Carbon nanoparticle (CNs) sentinel lymph node mapping
- CNs Group: Adults with clinically node-negative papillary thyroid carcinoma (cN0-PTC) who undergo intraoperative sentinel lymph node mapping using carbon nanoparticles (CNs) alone.
  Intervention: 0.2 ml of carbon nanoparticle suspension (concentration: 50 mg/ml) injected at multiple points around the thyroid tumor under ultrasound guidance. Black staining is used to visualize lymph nodes during surgery.
  Participants undergo standard thyroid surgery including thyroid lobectomy and central lymph node dissection, with additional dissection based on intraoperative findings.
  Interventions: Diagnostic Test: Indocyanine green (ICG) sentinel lymph node mapping
- ICG+CNs Group (Dual-Tracer): Adults with clinically node-negative papillary thyroid carcinoma (cN0-PTC) who undergo intraoperative sentinel lymph node mapping using combined indocyanine green and carbon nanoparticles (dual-tracer technique).
  Intervention: A mixture of 0.1 ml ICG solution (concentration: 2.5 mg/ml) and 0.1 ml carbon nanoparticle suspension (concentration: 50 mg/ml) injected at multiple points around the thyroid tumor under ultrasound guidance. Near-infrared fluorescence imaging combined with visual black staining is used to visualize lymphatic drainage and identify sentinel lymph nodes.
  This group also undergoes deep learning video analysis of the fluorescence imaging process to predict lymph node metastasis.
  Participants undergo standard thyroid surgery including thyroid lobectomy and central lymph node dissection, with additional dissection based on intraoperative findings.
  Interventions: Diagnostic Test: Dual-tracer (ICG combined with CNs) sentinel lymph node mapping

INTERVENTIONS:
Diagnostic Test: Indocyanine green (ICG) sentinel lymph node mapping — Intraoperative sentinel lymph node mapping using indocyanine green (ICG) with near-infrared fluorescence imaging.
  Preparation: ICG powder (25 mg) is dissolved in 10 ml sterile water to achieve a concentration of 2.5 mg/ml.
  Administration: 0.2 ml of ICG solution is injected at multiple points around the thyroid tumor under real-time ultrasound guidance using a precision multi-point stereotactic injection technique.
  Visualization: A near-infrared fluorescence imaging system (excitation wavelength 750-800 nm, emission wavelength 820 nm) is used to visualize lymphatic channels and identify sentinel lymph nodes in real time during surgery.
  The sentinel lymph node is defined as the first lymph node that shows fluorescence signal after tracer injection.
  Other Names: ICG fluorescence lymphography; Near-infrared fluorescence sentinel lymph node identification
  Groups: CNs Group
Diagnostic Test: Carbon nanoparticle (CNs) sentinel lymph node mapping — Intraoperative sentinel lymph node mapping using carbon nanoparticle suspension with visual identification.
  Preparation: Carbon nanoparticle suspension is used at the commercial concentration of 50 mg/ml.
  Administration: 0.2 ml of carbon nanoparticle suspension is injected at multiple points around the thyroid tumor under real-time ultrasound guidance using a precision multi-point stereotactic injection technique.
  Visualization: Carbon nanoparticles (diameter 150 nm) selectively enter lymphatic channels and accumulate in lymph nodes, producing visible black staining. Surgeons identify sentinel lymph nodes by direct visual inspection of black-stained nodes.
  The sentinel lymph node is defined as the first lymph node that shows black staining after tracer injection.
  Other Names: Carbon nanoparticle suspension lymph node tracing; Nano-carbon lymphatic mapping
  Groups: ICG Group
Diagnostic Test: Dual-tracer (ICG combined with CNs) sentinel lymph node mapping — Intraoperative sentinel lymph node mapping using combined indocyanine green and carbon nanoparticles with near-infrared fluorescence imaging and visual identification.
  Preparation: 0.1 ml of ICG solution (2.5 mg/ml) is mixed with 0.1 ml of carbon nanoparticle suspension (50 mg/ml) to form a 0.2 ml dual-tracer composite agent.
  Administration: The mixed tracer is injected at multiple points around the thyroid tumor under real-time ultrasound guidance using a precision multi-point stereotactic injection technique.
  Visualization: Near-infrared fluorescence imaging captures real-time lymphatic flow dynamics (ICG component), while black staining provides durable visual lymph node identification (CNs component). Video recording documents the entire sentinel lymph node visualization process for at least 5 minutes at 1920x1080 resolution.
  Deep learning analysis: In this group, video recordings are analyzed using nine deep learning models to extract spatiotemporal features and predict second
  Other Names: Combined ICG and carbon nanoparticle lymphatic mapping; Dual-tracer fluorescence and visual lymph node identification
  Groups: ICG+CNs Group (Dual-Tracer)

SUMMARY:
The goal of this observational study is to learn if a computer program (deep learning) can accurately predict lymph node spread in adults with papillary thyroid cancer who have no signs of lymph node involvement before surgery (called cN0). The main questions it aims to answer are:

* Can video analysis of lymph node mapping during surgery predict if cancer has spread to lymph nodes beyond the first-draining (sentinel) lymph node?
* Can this prediction help surgeons decide how much tissue to remove during surgery?

During surgery, participants will receive an injection of two special dyes (carbon nanoparticles and indocyanine green) near the thyroid tumor. These dyes travel through the lymphatic system and help surgeons see the lymph nodes. A special camera records a video of how the dyes move and light up the lymph nodes.

Researchers will use computer programs to analyze these videos along with other medical information (such as ultrasound results and tumor characteristics) to predict whether cancer has spread to additional lymph nodes. The predictions will be compared against the actual results from tissue samples examined after surgery.

Participants will receive standard thyroid cancer surgery. The study does not change the surgical treatment. The video recording adds no extra risk to participants.

DETAILED DESCRIPTION:
BACKGROUND AND RATIONALE:

Papillary thyroid carcinoma (PTC) is one of the fastest-growing cancers worldwide. A major challenge in treating PTC is that 30% to 80% of patients who appear to have no lymph node involvement before surgery (clinically node-negative, or cN0) actually have hidden (occult) cancer spread to their lymph nodes. Current imaging methods like ultrasound often miss these small areas of cancer spread.

This creates a difficult decision for surgeons: removing too many lymph nodes increases the risk of complications such as damage to the parathyroid glands (which control calcium levels) and the nerves that control the voice. However, removing too few lymph nodes may leave cancer behind, which can lead to recurrence.

Sentinel lymph node (SLN) mapping is a technique that identifies the first lymph nodes that drain from a tumor. The idea is that if cancer spreads through the lymphatic system, it will reach these sentinel nodes first. However, current single-tracer methods for SLN mapping in thyroid cancer have limitations and variable results.

This study uses a dual-tracer approach that combines two different dyes:

1. Carbon nanoparticles (CNs): These provide long-lasting black staining that helps surgeons see lymph nodes clearly
2. Indocyanine green (ICG): This dye glows under near-infrared light, allowing real-time visualization of lymphatic flow

By combining these two tracers, surgeons can see both the structure of lymph nodes and how lymphatic fluid flows through them over time.

STUDY DESIGN:

This is a prospective, single-center, observational cohort study. The study does not change the surgical treatment that participants receive. All participants undergo standard thyroid cancer surgery with lymph node removal as determined by their surgical team.

STUDY PROCEDURES:

1. Pre-operative Assessment:

   All participants undergo standard pre-operative evaluation including:
   * Physical examination
   * Thyroid ultrasound with detailed lymph node assessment
   * Fine-needle aspiration biopsy to confirm PTC diagnosis
   * Genetic testing for common mutations (such as BRAF)
   * Standard blood tests
2. Surgical Procedure:

   During surgery, participants receive the dual-tracer injection under ultrasound guidance. The injection is given at multiple points around the thyroid tumor. The specific preparation is:
   * 0.1 ml of ICG solution (concentration: 2.5 mg/ml)
   * 0.1 ml of carbon nanoparticle suspension (concentration: 50 mg/ml) These are mixed together and injected using precise, multi-point technique.
3. Video Recording:

   A near-infrared fluorescence imaging system records the entire process of lymph node visualization. The recording captures:
   * How the dyes spread through the lymphatic channels
   * When each lymph node first becomes visible
   * How the fluorescence signal changes over time
   * The pattern of lymphatic drainage

   Videos are recorded at high resolution (1920 × 1080 pixels) at approximately 30 frames per second. A standardized 3-minute segment is extracted from each video for analysis, providing 150 frames per patient.
4. Surgical Decisions:

   The sentinel lymph node (the first node that lights up) is removed and sent for immediate frozen section analysis. Based on standard criteria, surgeons decide whether to perform:
   * Ipsilateral central lymph node dissection (removing lymph nodes on the same side as the tumor)
   * Lateral lymph node dissection (if certain criteria are met)
   * Contralateral central dissection (removing lymph nodes on the opposite side)

   These decisions follow the standard surgical protocol at our institution and are not influenced by the deep learning predictions.
5. Pathological Examination:

All removed lymph nodes are examined by pathologists to determine:

* Whether the sentinel lymph node contains cancer (SLNM status)
* Whether second-echelon lymph nodes contain cancer (SeLNM)
* Whether non-sentinel lymph nodes contain cancer (NsLNM)
* The number and location of all positive lymph nodes

DATA COLLECTION AND ANALYSIS:

Clinical Data (32 variables):

* Demographics: age, sex, body mass index
* Ultrasound features: tumor size, location, margins, calcification patterns, aspect ratio, TI-RADS classification
* Pathological features: multifocality, extrathyroidal extension, capsular invasion
* Genetic data: BRAF mutation status and other relevant mutations

Video Analysis:

Two experienced surgeons (each with more than 10 years of experience) manually identify and outline the regions of interest (the sentinel lymph nodes) in each video frame. This creates 19,650 mask images across all participants.

Feature Extraction:

The deep learning system extracts multiple types of features:

Spatial Features (2,048 dimensions):

* Image features from a pre-trained neural network (EfficientNet-B5)
* Grayscale characteristics
* Shape and morphological features
* Hu moment descriptors (mathematical descriptions of shape)

Temporal Features (20 dimensions):

* Frame-to-frame differences showing how the image changes
* Optical flow measurements showing movement patterns
* Fluorescence intensity changes over time
* Flow velocity measurements at specific time points

DEEP LEARNING MODELS:

Nine different deep learning architectures are developed and compared:

1. Convolutional Neural Network (CNN): Extracts local spatial features from images
2. Long Short-Term Memory (LSTM): Captures patterns in time-series data
3. CNN + LSTM: Combines spatial and temporal feature extraction
4. CNN + LSTM + Attention: Adds attention mechanism to focus on important time points
5. Transformer: Uses self-attention to capture global patterns in sequential data
6. Crossformer: A specialized architecture for time-series analysis
7. 3D-CNN: Processes video data as three-dimensional volumes
8. LSTM + Transformer: Hybrid model combining LSTM and Transformer strengths
9. LSTM + Crossformer: Hybrid model combining LSTM and Crossformer

All models use:

* Binary cross-entropy loss function
* Adam optimizer for training
* Data augmentation (rotation, scaling, noise injection) to prevent overfitting
* Weighted loss functions to handle class imbalance
* Dropout regularization

MODEL EVALUATION:

Models are evaluated using 10-fold stratified cross-validation, ensuring balanced distribution of outcomes in training and testing sets. Performance metrics include:

* Area Under the ROC Curve (AUC): Measures overall discrimination ability
* Accuracy: Percentage of correct predictions
* Sensitivity: Ability to correctly identify patients with metastasis
* Specificity: Ability to correctly identify patients without metastasis
* Positive Predictive Value: Probability that a positive prediction is correct
* Negative Predictive Value: Probability that a negative prediction is correct
* F1 Score: Balance between precision and recall
* Brier Score: Calibration of predicted probabilities

Additional analyses include:

* Decision curve analysis to assess clinical utility
* Calibration curves to check prediction reliability
* Learning curves to assess overfitting
* DeLong test for statistical comparison between models
* Probability-based model ranking approach (PMRA)

MODEL INTERPRETABILITY:

To understand how the model makes predictions, we use SHapley Additive exPlanations (SHAP) analysis. This technique:

* Identifies which features contribute most to predictions
* Shows how each feature affects individual predictions
* Reveals whether the model relies on clinically meaningful factors
* Provides transparency into the "black box" of deep learning

OUTCOMES:

Primary Outcomes:

1. Second-echelon lymph node metastasis (SeLNM): Cancer spread to lymph nodes beyond the sentinel node in the drainage pathway
2. Non-sentinel lymph node metastasis (NsLNM): Cancer spread to any lymph node other than the sentinel node

Both outcomes are determined by final pathological examination of surgically removed tissue (the gold standard).

Secondary Outcomes:

* Model performance metrics (AUC, sensitivity, specificity, etc.)
* Feature importance rankings from SHAP analysis
* Comparison of model architectures

STATISTICAL CONSIDERATIONS:

Sample Size:

Based on power calculations assuming:

* Alpha = 0.05 (significance level)
* Power = 0.80
* Expected sensitivity difference of 20% between methods
* Expected prevalence of lymph node metastasis of 50%

A minimum of 335 participants was calculated. Due to strict inclusion criteria and video quality requirements, 131 participants with complete, high-quality data were included in the final analysis.

Statistical Methods:

* Descriptive statistics for baseline characteristics
* Chi-square or Fisher exact test for categorical variables
* Mann-Whitney U test for continuous variables
* DeLong test for comparing AUC values between models
* 95% confidence intervals for all performance metrics

FOLLOW-UP:

While the primary analysis focuses on intraoperative prediction, participants are followed according to standard clinical care protocols. Long-term outcomes including recurrence-free survival may be analyzed in future studies.

ETHICAL CONSIDERATIONS:

This study was approved by the Ethics Committee of the First Affiliated Hospital of Chongqing Medical University (Approval No. 2023-322). All participants provided written informed consent before enrollment.

The study poses minimal additional risk to participants because:

* The dual-tracer injection uses agents already approved for clinical use
* The video recording is non-invasive and does not affect surgical decisions
* All surgical decisions are made according to standard protocols
* The deep learning analysis is performed retrospectively and does not influence treatment

POTENTIAL IMPACT:

If successful, this approach could:

1. Help surgeons make more informed decisions about the extent of lymph node removal
2. Reduce unnecessary extensive surgery in low-risk patients
3. Ensure adequate surgery in high-risk patients who might otherwise be undertreated
4. Provide real-time, objective decision support during surgery
5. Standardize the interpretation of lymphatic mapping across different surgeons and centers
6. Serve as a training tool for less experienced surgeons

LIMITATIONS:

* Single-center study, which may limit generalizability
* Relatively small sample size due to strict quality requirements
* Manual annotation of regions of interest may introduce variability
* Deep learning models require validation in external cohorts
* Real-time implementation during surgery requires further development

FUTURE DIRECTIONS:

* External validation in multiple centers
* Development of real-time prediction software for intraoperative use
* Integration with other imaging modalities
* Prospective interventional trials to assess clinical benefit of AI-guided surgery

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older at the time of enrollment
2. Histologically confirmed papillary thyroid carcinoma (PTC) by preoperative fine-needle aspiration biopsy
3. Clinically node-negative (cN0) status confirmed by preoperative imaging (ultrasound and/or cross-sectional imaging showing no evidence of lymph node metastasis)
4. Scheduled to undergo thyroid surgery with simultaneous central lymph node dissection
5. Willing and able to provide written informed consent
6. Complete preoperative clinical data available, including:

   * Demographic information (age, sex, body mass index)
   * Thyroid ultrasound report with detailed tumor characteristics
   * Fine-needle aspiration biopsy pathology report
   * Genetic testing results (when available)
7. Able to undergo intraoperative dual-tracer sentinel lymph node mapping with near-infrared fluorescence video recording

Exclusion Criteria:

1. History of previous neck surgery (including thyroid surgery, parathyroid surgery, or other cervical operations)
2. History of external beam radiotherapy to the head and neck region
3. Diagnosis of thyroid malignancy other than papillary thyroid carcinoma (e.g., follicular thyroid carcinoma, medullary thyroid carcinoma, anaplastic thyroid carcinoma, or thyroid lymphoma)
4. Known allergy or hypersensitivity to indocyanine green (ICG), iodine, or carbon nanoparticles
5. Severe hepatic insufficiency (ICG is metabolized by the liver)
6. Pregnancy or breastfeeding
7. Incomplete medical records or missing essential preoperative data
8. Refusal to undergo dual-tracer imaging procedure
9. Inability to obtain satisfactory intraoperative near-infrared fluorescence video recording due to technical issues or poor image quality
10. Participation in another interventional clinical trial that may interfere with the current study
11. Any condition that, in the investigator's opinion, would compromise the participant's safety or the quality of the study data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults diagnosed with clinically node-negative papillary thyroid carcinoma (cN0-PTC) who are scheduled to undergo surgical treatment at the Department of Breast and Thyroid Surgery, First Affiliated Hospital of Chongqing Medical University, Chongqing, China. Participants are identified through routine clinical care and preoperative evaluation. The study population includes patients with primary PTC confirmed by fine-needle aspiration biopsy who have no evidence of lymph node metastasis on preoperative ultrasound or other imaging studies. Both male and female adults aged 18 years and older are eligible regardless of tumor size, location, or genetic mutation status.
Sampling Method: Non-Probability Sample
Enrollment: 131 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Sentinel Lymph Node Metastasis (SLNM) Status | immediately after the surgery
  The presence or absence of cancer metastasis in the sentinel lymph node, determined by postoperative histopathological examination (paraffin section) as the gold standard. SLNM is classified as positive (macrometastasis or micrometastasis present) or negative (no metastasis). The SLNM rate is calculated as: number of participants with positive sentinel lymph nodes divided by total number of participants with successfully identified sentinel lymph nodes.
Sentinel Lymph Node Detection Rate | immediately after the surgery
  The proportion of participants in whom sentinel lymph nodes are successfully identified using each tracer method (ICG alone, CNs alone, or ICG+CNs dual-tracer). A sentinel lymph node is defined as the first lymph node visualized after tracer injection. Detection rate is calculated as: number of participants with successfully identified sentinel lymph nodes divided by total number of participants in each group, expressed as a percentage.
Second-Echelon Lymph Node Metastasis (SeLNM) | perioperatively
  The presence or absence of cancer metastasis in second-echelon lymph nodes (lymph nodes beyond the sentinel node in the lymphatic drainage pathway), determined by postoperative histopathological examination. SeLNM is the primary prediction target for the deep learning models in the ICG+CNs group. SeLNM status is classified as positive or negative based on paraffin section pathology results.
Non-Sentinel Lymph Node Metastasis (NsLNM) | perioperatively
  The presence or absence of cancer metastasis in any lymph node other than the sentinel lymph node, determined by postoperative histopathological examination. NsLNM includes metastasis in central compartment nodes (prelaryngeal, pretracheal, paratracheal, and nodes posterior to recurrent laryngeal nerve) and lateral compartment nodes when dissected. NsLNM is the second primary prediction target for the deep learning models in the ICG+CNs group.

SECONDARY OUTCOMES:
Sensitivity of Sentinel Lymph Node Mapping | through study completion, an average of 1 year
  The ability of each tracer method to correctly identify participants who have lymph node metastasis. Sensitivity is calculated as: true positives divided by (true positives + false negatives), expressed as a percentage. A true positive is defined as a positive sentinel lymph node in a participant with confirmed central lymph node metastasis on final pathology. Compared among ICG, CNs, and ICG+CNs groups.
Specificity of Sentinel Lymph Node Mapping | through study completion, an average of 1 year
  The ability of each tracer method to correctly identify participants who do not have lymph node metastasis. Specificity is calculated as: true negatives divided by (true negatives + false positives), expressed as a percentage. A true negative is defined as a negative sentinel lymph node in a participant with no central lymph node metastasis on final pathology. Compared among ICG, CNs, and ICG+CNs groups.
Positive Predictive Value (PPV) of Sentinel Lymph Node Mapping | through study completion, an average of 1 year
  The probability that participants with a positive sentinel lymph node truly have central lymph node metastasis. PPV is calculated as: true positives divided by (true positives + false positives), expressed as a percentage. Compared among ICG, CNs, and ICG+CNs groups.
Negative Predictive Value (NPV) of Sentinel Lymph Node Mapping | through study completion, an average of 1 year
  The probability that participants with a negative sentinel lymph node truly do not have central lymph node metastasis. NPV is calculated as: true negatives divided by (true negatives + false negatives), expressed as a percentage. A high NPV indicates that a negative sentinel lymph node reliably rules out metastatic disease. Compared among ICG, CNs, and ICG+CNs groups.
Deep Learning Model Performance - Area Under ROC Curve (AUC) | through study completion, an average of 1 year
  The area under the receiver operating characteristic curve for each deep learning model (CNN, LSTM, CNN+LSTM, CNN+LSTM+Attention, Transformer, Crossformer, 3D-CNN, LSTM+Transformer, LSTM+Crossformer) in predicting SeLNM and NsLNM in the ICG+CNs group. AUC ranges from 0 to 1, with higher values indicating better discrimination. Evaluated using 10-fold stratified cross-validation.
Deep Learning Model Performance - Accuracy, Sensitivity, and Specificity | through study completion, an average of 1 year
  Performance metrics of the optimal deep learning model for predicting SeLNM and NsLNM in the ICG+CNs group. Accuracy is the proportion of correct predictions. Sensitivity is the proportion of actual positive cases correctly identified. Specificity is the proportion of actual negative cases correctly identified. All metrics expressed as percentages with 95% confidence intervals.

OTHER OUTCOMES:
Number of Sentinel Lymph Nodes Identified | immediately after surgery
  The mean number of sentinel lymph nodes identified per participant using each tracer method. Compared among ICG, CNs, and ICG+CNs groups using appropriate statistical tests.
Total Number of Lymph Nodes Retrieved | perioperatively
  The total number of lymph nodes retrieved during central and lateral lymph node dissection per participant. Reported as mean with standard deviation for each group.
Feature Importance from SHAP Analysis | through study completion, an average of 1 year
  Identification and ranking of the most important predictive features contributing to the deep learning model predictions, determined by SHapley Additive exPlanations (SHAP) analysis. Features include temporal fluorescence-flow characteristics, spatial structural features, and clinical variables. Reported as mean absolute SHAP values for top contributing features.
Surgical Complications | up to 24 weeks
  Incidence of surgery-related complications including: transient or permanent hypoparathyroidism (based on postoperative calcium and parathyroid hormone levels), transient or permanent recurrent laryngeal nerve injury (based on postoperative laryngoscopy), postoperative bleeding requiring intervention, and wound infection. Reported as number and percentage of participants in each group.
Tracer-Related Adverse Events | perioperatively
  Incidence of adverse events related to tracer injection, including allergic reactions, injection site reactions, and any other tracer-associated complications. ICG-related adverse events are expected to be less than 0.05% based on published literature. Reported as number and percentage of participants in each group.

CONTACTS AND LOCATIONS:
Overall Officials: Xinliang Su, MD,PhD, Study Director — First Affiliated Hospital of Chongqing Medical University; Han Gao, MD,PhD, Study Chair — Women and Children's Hospital of Chongqing Medical University; Xinliang Su, MD,PhD, Principal Investigator — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, China

IPD SHARING:
Plan to Share IPD: Undecided
A decision regarding individual participant data sharing has not yet been finalized. The study team is currently evaluating:
  1. Technical feasibility of de-identifying video-based imaging data
  2. Institutional and ethical requirements for data sharing
  3. Development of appropriate data use agreements
  The IPD sharing plan will be updated prior to publication of the primary study results. Interested researchers may contact the Principal Investigator (suxinliang@21cn.com) to discuss potential future data access.

REFERENCES:
- [Result] Qian T, Zhou Y, Yao J, Ni C, Asif S, Chen C, Lv L, Ou D, Xu D. Deep learning based analysis of dynamic video ultrasonography for predicting cervical lymph node metastasis in papillary thyroid carcinoma. Endocrine. 2025 Mar;87(3):1060-1069. doi: 10.1007/s12020-024-04091-w. Epub 2024 Nov 18. PMID 39556263
- [Result] Ding X, Liu Y, Zhao J, Wang R, Li C, Luo Q, Shen C. A novel wavelet-transform-based convolution classification network for cervical lymph node metastasis of papillary thyroid carcinoma in ultrasound images. Comput Med Imaging Graph. 2023 Oct;109:102298. doi: 10.1016/j.compmedimag.2023.102298. Epub 2023 Sep 9. PMID 37769402
- [Result] Yang D, Li T, Li L, Chen S, Li X. Multi-modal convolutional neural network-based thyroid cytology classification and diagnosis. Hum Pathol. 2025 Jul;161:105868. doi: 10.1016/j.humpath.2025.105868. Epub 2025 Jul 4. PMID 40617519
- [Result] Chu X, Wang T, Chen M, Li J, Wang L, Wang C, Wang H, Wong ST, Chen Y, Li H. Deep learning model for malignancy prediction of TI-RADS 4 thyroid nodules with high-risk characteristics using multimodal ultrasound: A multicentre study. Comput Med Imaging Graph. 2025 Sep;124:102576. doi: 10.1016/j.compmedimag.2025.102576. Epub 2025 May 26. PMID 40446583
- [Result] Liang M, Zhu T, Huang N, Zhang L, Yang C, Gao H, Zhang X, Li P, Cheng M, Wang K. Incorporating sentinel chain involvement pattern to predict non-sentinel lymph nodes status in breast cancer after neoadjuvant chemotherapy. Clin Transl Oncol. 2026 Jan;28(1):203-214. doi: 10.1007/s12094-025-03993-z. Epub 2025 Jul 31. PMID 40745244
- [Result] Mittendorf EA, Hunt KK, Boughey JC, Bassett R, Degnim AC, Harrell R, Yi M, Meric-Bernstam F, Ross MI, Babiera GV, Kuerer HM, Hwang RF. Incorporation of sentinel lymph node metastasis size into a nomogram predicting nonsentinel lymph node involvement in breast cancer patients with a positive sentinel lymph node. Ann Surg. 2012 Jan;255(1):109-15. doi: 10.1097/SLA.0b013e318238f461. PMID 22167004
- [Result] Zhou L, Yao J, Ou D, Li M, Lei Z, Wang L, Xu D. A multi-institutional study of association of sonographic characteristics with cervical lymph node metastasis in unifocal papillary thyroid carcinoma. Front Endocrinol (Lausanne). 2022 Sep 23;13:965241. doi: 10.3389/fendo.2022.965241. eCollection 2022. PMID 36213266
- [Result] Khan SU, Fatima K, Malik F, Kalkavan H, Wani A. Cancer metastasis: Molecular mechanisms and clinical perspectives. Pharmacol Ther. 2023 Oct;250:108522. doi: 10.1016/j.pharmthera.2023.108522. Epub 2023 Sep 1. PMID 37661054
- [Result] Cao R, Ji H, Feng N, Zhang Y, Yang X, Andersson P, Sun Y, Tritsaris K, Hansen AJ, Dissing S, Cao Y. Collaborative interplay between FGF-2 and VEGF-C promotes lymphangiogenesis and metastasis. Proc Natl Acad Sci U S A. 2012 Sep 25;109(39):15894-9. doi: 10.1073/pnas.1208324109. Epub 2012 Sep 11. PMID 22967508
- [Result] Li Y, Chen H, Zhao Y, Yan Q, Chen L, Song Q. circUBE2G1 interacts with hnRNPU to promote VEGF-C-mediated lymph node metastasis of lung adenocarcinoma. Front Oncol. 2024 Nov 27;14:1455909. doi: 10.3389/fonc.2024.1455909. eCollection 2024. PMID 39664183
- [Result] Guang Y, Wan F, He W, Zhang W, Gan C, Dong P, Zhang H, Zhang Y. A model for predicting lymph node metastasis of thyroid carcinoma: a multimodality convolutional neural network study. Quant Imaging Med Surg. 2023 Dec 1;13(12):8370-8382. doi: 10.21037/qims-23-318. Epub 2023 Nov 7. PMID 38106318
- [Result] Luo QW, Gao S, Lv X, Li SJ, Wang BF, Han QQ, Wang YP, Guan QL, Gong T. A novel tool for predicting the risk of central lymph node metastasis in patients with papillary thyroid microcarcinoma: a retrospective cohort study. BMC Cancer. 2022 Jun 2;22(1):606. doi: 10.1186/s12885-022-09655-5. PMID 35655253
- [Result] Popadich A, Levin O, Lee JC, Smooke-Praw S, Ro K, Fazel M, Arora A, Tolley NS, Palazzo F, Learoyd DL, Sidhu S, Delbridge L, Sywak M, Yeh MW. A multicenter cohort study of total thyroidectomy and routine central lymph node dissection for cN0 papillary thyroid cancer. Surgery. 2011 Dec;150(6):1048-57. doi: 10.1016/j.surg.2011.09.003. PMID 22136820
- [Result] Huang C, Cong S, Shang S, Wang M, Zheng H, Wu S, An X, Liang Z, Zhang B. Web-Based Ultrasonic Nomogram Predicts Preoperative Central Lymph Node Metastasis of cN0 Papillary Thyroid Microcarcinoma. Front Endocrinol (Lausanne). 2021 Sep 7;12:734900. doi: 10.3389/fendo.2021.734900. eCollection 2021. PMID 34557165
- [Result] Wang Y, Deng C, Shu X, Yu P, Wang H, Su X, Tan J. Risk Factors and a Prediction Model of Lateral Lymph Node Metastasis in CN0 Papillary Thyroid Carcinoma Patients With 1-2 Central Lymph Node Metastases. Front Endocrinol (Lausanne). 2021 Oct 15;12:716728. doi: 10.3389/fendo.2021.716728. eCollection 2021. PMID 34721289
- [Result] Chun L, Wang D, He L, Li D, Fu Z, Xue S, Su X, Zhou J. Explainable machine learning model for predicting paratracheal lymph node metastasis in cN0 papillary thyroid cancer. Sci Rep. 2024 Sep 27;14(1):22361. doi: 10.1038/s41598-024-73837-3. PMID 39333646
- [Result] Du W, Fang Q, Zhang X, Dai L. Metastasis of cN0 Papillary Thyroid Carcinoma of the Isthmus to the Lymph Node Posterior to the Right Recurrent Laryngeal Nerve. Front Endocrinol (Lausanne). 2021 May 10;12:677986. doi: 10.3389/fendo.2021.677986. eCollection 2021. PMID 34040587
- [Result] He F, Chen S, Liu X, Yang X, Qin X. Multimodal Deep Learning Model Based on Ultrasound and Cytological Images Predicts Risk Stratification of cN0 Papillary Thyroid Carcinoma. Acad Radiol. 2025 Sep;32(9):5091-5099. doi: 10.1016/j.acra.2025.06.043. Epub 2025 Jul 14. PMID 40664556
- [Result] Yin SM, Lien JJ, Chiu IM. Deep learning implementation for extrahepatic bile duct detection during indocyanine green fluorescence-guided laparoscopic cholecystectomy: pilot study. BJS Open. 2025 Mar 4;9(2):zraf013. doi: 10.1093/bjsopen/zraf013. PMID 40119711
- [Result] Shen B, Zhang Z, Shi X, Cao C, Zhang Z, Hu Z, Ji N, Tian J. Real-time intraoperative glioma diagnosis using fluorescence imaging and deep convolutional neural networks. Eur J Nucl Med Mol Imaging. 2021 Oct;48(11):3482-3492. doi: 10.1007/s00259-021-05326-y. Epub 2021 Apr 27. PMID 33904984
- [Result] Chang YY, Yang HP, Chen YY, Yen HH. Comparison of the performance between an AI-based vision transformer and human endoscopists in predicting the endoscopic and histologic activities of ulcerative colitis. Digit Health. 2026 Jan 5;12:20552076251412694. doi: 10.1177/20552076251412694. eCollection 2026 Jan-Dec. PMID 41509873
- [Result] Kumar R, Sethia K, Kumar V. Video-endoscopic versus open inguinal lymphadenectomy: Long-term oncological outcomes in penile cancer. BJUI Compass. 2026 Jan 6;7(1):e70153. doi: 10.1002/bco2.70153. eCollection 2026 Jan. PMID 41509534
- [Result] Oh N, Kim B, Kim T, Rhu J, Kim J, Choi GS. Real-time segmentation of biliary structure in pure laparoscopic donor hepatectomy. Sci Rep. 2024 Sep 28;14(1):22508. doi: 10.1038/s41598-024-73434-4. PMID 39341910
- [Result] Jha D, Ali S, Tomar NK, Johansen HD, Johansen D, Rittscher J, Riegler MA, Halvorsen P. Real-Time Polyp Detection, Localization and Segmentation in Colonoscopy Using Deep Learning. IEEE Access. 2021 Mar 4;9:40496-40510. doi: 10.1109/ACCESS.2021.3063716. eCollection 2021. PMID 33747684
- [Result] Dolidze DD, Shabunin AV, Mumladze RB, Vardanyan AV, Covantsev SD, Shulutko AM, Semikov VI, Isaev KM, Kazaryan AM. A Narrative Review of Preventive Central Lymph Node Dissection in Patients With Papillary Thyroid Cancer - A Necessity or an Excess. Front Oncol. 2022 Jun 29;12:906695. doi: 10.3389/fonc.2022.906695. eCollection 2022. PMID 35847927
- [Result] Giordano D, Valcavi R, Thompson GB, Pedroni C, Renna L, Gradoni P, Barbieri V. Complications of central neck dissection in patients with papillary thyroid carcinoma: results of a study on 1087 patients and review of the literature. Thyroid. 2012 Sep;22(9):911-7. doi: 10.1089/thy.2012.0011. Epub 2012 Jul 24. PMID 22827494
- [Result] Zhang L, Cheng M, Lin Y, Zhang J, Shen B, Chen Y, Yang C, Yang M, Zhu T, Gao H, Ji F, Li J, Wang K. Ultrasound-assisted carbon nanoparticle suspension mapping versus dual tracer-guided sentinel lymph node biopsy in patients with early breast cancer (ultraCars): phase III randomized clinical trial. Br J Surg. 2022 Nov 22;109(12):1232-1238. doi: 10.1093/bjs/znac311. PMID 36074703
- [Result] Bargon CA, Huibers A, Young-Afat DA, Jansen BAM, Borel-Rinkes IHM, Lavalaye J, van Slooten HJ, Verkooijen HM, van Swol CFP, Doeksen A. Sentinel Lymph Node Mapping in Breast Cancer Patients Through Fluorescent Imaging Using Indocyanine Green: The INFLUENCE Trial. Ann Surg. 2022 Nov 1;276(5):913-920. doi: 10.1097/SLA.0000000000005633. Epub 2022 Jul 27. PMID 35894448
- [Result] Solis O, Addae J, Sweeting R, Meszoely I, Grau A, Kauffmann R, Kelley M, McCaffrey R, Hewitt K. Cost containment analysis of superparamagnetic iron oxide (SPIO) injection in patients with ductal carcinoma in situ. Breast Cancer Res Treat. 2024 Dec;208(3):565-568. doi: 10.1007/s10549-024-07451-2. Epub 2024 Aug 1. PMID 39085674
- [Result] Madadi M, Khoee S. Magnetite-based Janus nanoparticles, their synthesis and biomedical applications. Wiley Interdiscip Rev Nanomed Nanobiotechnol. 2023 Nov-Dec;15(6):e1908. doi: 10.1002/wnan.1908. Epub 2023 Jun 4. PMID 37271573
- [Result] Marengo M, Martin CJ, Rubow S, Sera T, Amador Z, Torres L. Radiation Safety and Accidental Radiation Exposures in Nuclear Medicine. Semin Nucl Med. 2022 Mar;52(2):94-113. doi: 10.1053/j.semnuclmed.2021.11.006. Epub 2021 Dec 13. PMID 34916044
- [Result] Garau LM, Rubello D, Ferretti A, Boni G, Volterrani D, Manca G. Sentinel lymph node biopsy in small papillary thyroid cancer. A review on novel surgical techniques. Endocrine. 2018 Nov;62(2):340-350. doi: 10.1007/s12020-018-1658-5. Epub 2018 Jul 2. PMID 29968226
- [Result] Garau LM, Rubello D, Morganti R, Boni G, Volterrani D, Colletti PM, Manca G. Sentinel Lymph Node Biopsy in Small Papillary Thyroid Cancer: A Meta-analysis. Clin Nucl Med. 2019 Feb;44(2):107-118. doi: 10.1097/RLU.0000000000002378. PMID 30418209
- [Result] Santrac N, Markovic I, Medic Milijic N, Goran M, Buta M, Djurisic I, Dzodic R. Sentinel lymph node biopsy in medullary thyroid microcarcinomas. Endocr J. 2020 Mar 28;67(3):295-304. doi: 10.1507/endocrj.EJ19-0409. Epub 2019 Dec 3. PMID 31801918
- [Result] Boschin IM, Bertazza L, Scaroni C, Mian C, Pelizzo MR. Sentinel lymph node mapping: current applications and future perspectives in thyroid carcinoma. Front Med (Lausanne). 2023 Oct 24;10:1231566. doi: 10.3389/fmed.2023.1231566. eCollection 2023. PMID 37942415
- [Result] Likhterov I, Reis LL, Urken ML. Central compartment management in patients with papillary thyroid cancer presenting with metastatic disease to the lateral neck: Anatomic pathways of lymphatic spread. Head Neck. 2017 May;39(5):853-859. doi: 10.1002/hed.24568. Epub 2017 Mar 2. PMID 28252836
- [Result] Lopez-Martinez R. [Immunological characteristics in candidiasis]. Prensa Med Mex. 1974 Nov-Dec;39(11-12):468-71. No abstract available. Spanish. PMID 4457868
- [Result] Flagiello D, Gibaud A, Dutrillaux B, Poupon MF, Malfoy B. Distinct patterns of all-trans retinoic acid dependent expression of HOXB and HOXC homeogenes in human embryonal and small-cell lung carcinoma cell lines. FEBS Lett. 1997 Oct 6;415(3):263-7. doi: 10.1016/s0014-5793(97)01118-6. PMID 9357979
- [Result] Galili U. Evolution of alpha 1,3galactosyltransferase and of the alpha-Gal epitope. Subcell Biochem. 1999;32:1-23. doi: 10.1007/978-1-4615-4771-6_1. No abstract available. PMID 10391989
- [Result] Dogan H, Tasman F, Cehreli ZC. Effect of gutta-percha solvents at different temperatures on the calcium, phosphorus and magnesium levels of human root dentin. J Oral Rehabil. 2001 Aug;28(8):792-6. doi: 10.1046/j.1365-2842.2001.00714.x. PMID 11556962
- [Result] Izumi AK, Dawson KL. Zabon phytophotodermatitis: first case reports due to Citrus maxima. J Am Acad Dermatol. 2002 May;46(5 Suppl):S146-7. doi: 10.1067/mjd.2002.107489. PMID 12004296
- [Result] Chapchal G. [On the conservative therapy of joint contractures in hemophilia]. Schweiz Med Wochenschr. 1967 Jun 17;97(24):788-90. No abstract available. German. PMID 5593627
- [Result] Hardaway BW, Hoffer FA, Rao BN. Needle localization of small pediatric tumors for surgical biopsy. Pediatr Radiol. 2000 May;30(5):318-22. doi: 10.1007/s002470050748. PMID 10836594
- [Result] Sokoloff MH, Chung LW. Targeting angiogenic pathways involving tumor-stromal interaction to treat advanced human prostate cancer. Cancer Metastasis Rev. 1998-1999;17(4):307-15. doi: 10.1023/a:1006170612253. PMID 10453273
- [Result] Roller RJ, Herold BC. Characterization of a BHK(TK-) cell clone resistant to postattachment entry by herpes simplex virus types 1 and 2. J Virol. 1997 Aug;71(8):5805-13. doi: 10.1128/JVI.71.8.5805-5813.1997. PMID 9223469
- [Result] Hansma HG, Clegg DO, Kokkoli E, Oroudjev E, Tirrell M. Analysis of matrix dynamics by atomic force microscopy. Methods Cell Biol. 2002;69:163-93. doi: 10.1016/s0091-679x(02)69012-0. No abstract available. PMID 12070991

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-09-23): https://cdn.clinicaltrials.gov/large-docs/14/NCT07391514/Prot_SAP_000.pdf
  • Informed Consent Form (2023-09-23): https://cdn.clinicaltrials.gov/large-docs/14/NCT07391514/ICF_001.pdf